CLINICAL TRIAL: NCT03096145
Title: Pilot Study Phase - Nonsmoker Interventions to Increase Use of Quitline Services Among Racially Diverse Low Income Smokers
Brief Title: Support Person Intervention to Promote a Smoking Helpline Among Under Resourced Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christi Patten, Professor of Psychology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-006338
Record Dates: First submitted 2017-03-25; First posted 2017-03-30 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Tobacco Cessation
Keywords: tobacco; quitlines; social support; mobile support
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Intervention (Experimental): Behavioral: telephone counseling 1 sessions, mobile texting, and health incentive
  Interventions: Behavioral: Telephone counseling 1 session; Behavioral: Mobile texting; Behavioral: Health incentive

INTERVENTIONS:
Behavioral: Telephone counseling 1 session — 1 call coaching session for nonsmokers that will be piloted and adapted in this study
Behavioral: Mobile texting — nonsmokers will receive 3-5 text messages for 4 weeks
Behavioral: Health incentive — Smokers receive a $25 gift card if they call the quitline

SUMMARY:
This pilot study is being done to adapt an effective 1 session phone coaching intervention for nonsmoking support persons to a low income population. This study will also pilot new intervention components including text messaging and health incentives. The goal of the intervention is for support persons to prompt their smoker to use quitline services. To see if these methods are effective, smokers in this study will be asked to complete assessments about their quit attempts and smoking status. The study will also evaluate if the smokers use quitline services or not. The preliminary findings will be used to provide data for an R01 NIH grant submission.

DETAILED DESCRIPTION:
This is a proposal to conduct a pilot study to adapt an effective 1 session phone coaching intervention for nonsmoking support persons to a low income population. The study will also pilot new intervention components including text messaging and health incentives. The goal of the intervention is for support persons to prompt their smoker to use quitline services. The study will also build on prior work by enrolling smokers for assessments of quit attempts and smoking abstinence. The study uses a non-randomized, single group design. Thirty nonsmoker-smoker dyads will be enrolled in three waves of 10 each. The nonsmokers will receive different intervention components depending on the time of their enrollment. Nonsmokers will complete assessments at baseline and at 1 month follow-up. Smokers will be enrolled for assessments only at baseline and 3 month follow-up. The vendor for the Minnesota state quitline, Alere Wellbeing Inc. (a sole subsidiary of Optum) will track if smokers use quitline services over 3 months of follow-up. The aims of this pilot study are to: (1) Assess the feasibility of enrolling low income, racially diverse nonsmoker-smoker dyads; (2) Adapt and refine the support person intervention components to a low income population with feedback from the nonsmoker participants; and (3) Assess the feasibility of obtaining assessments from the smokers on quit attempts and smoking abstinence outcomes. The preliminary findings will be used to provide data for an R01 NIH grant submission.

ELIGIBILITY:
Nonsmoker Inclusion Criteria:

* Minnesota resident
* 18 years of age or older
* Is a never smoker or former smoker (no cigarette smoking in past 6 months)
* Has a low income defined as receiving state funded health insurance including medical assistance (e.g., Medicaid) or MinnesotaCare
* Has access to a working cellular telephone with text messaging capabilities
* Has a mailing address/P.O. box
* Have regular contact with a current smoker is at least 18 years of age, resides in MN
* Provided verbal consent

Nonsmoker Exclusion Criteria:

* Their smoker does not provide written informed consent

Smoker Study Inclusion Criteria:

* Minnesota resident
* 18 years of age or older
* Has a low income defined as receiving state funded health insurance including medical assistance (e.g., Medicaid) or MinnesotaCare
* Has access to a working phone
* Has a mailing address/P.O. box
* Has smoked at least 1 cigarette in the past 30 days (to include both light/intermittent as well as daily/frequent smokers thus enhancing generalizability)
* Has not participated in a stop smoking program in the past 3 months including receiving pharmacotherapy for smoking cessation
* Provided written informed consent

Smoker Exclusion Criteria:

* Their nonsmoker does not provide verbal consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2019-08-24 (Actual)

PRIMARY OUTCOMES:
Number of low-income nonsmoker-smoker dyads at 1 month follow-up | 1 month
  feasibility of retaining low-income nonsmoker-smoker dyads at the 1 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Christi A Patten, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials